CLINICAL TRIAL: NCT06872333
Title: Allogeneic Hematopoietic Stem Cell Transplant for Patients With High Risk Hemoglobinopathies and Other Red Cell Transfusion Dependent Disorders
Brief Title: Allo HSCT for High Risk Hemoglobinopathies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024LS140
Record Dates: First submitted 2025-03-05; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Graft Failure; Sickle Cell Disease; Hemoglobinopathies
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinopathies | interventions — Alemtuzumab; Whole-Body Irradiation; Insulin Infusion Systems; thymoglobulin; fludarabine; Busulfan; Thiotepa; Cyclophosphamide; Mesna; Sirolimus; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): Arm A Matched sib regimen - Age 6 -55 (per physician preference for patients over 6) Campath/TBI
  Interventions: Drug: Alemtuzumab; Radiation: Total Body Irradiation; Biological: Cell Infusion; Drug: Sirolimus; Drug: Mycophenolate Mofetil
- Arm B (Experimental): Arm B Matched sib regimen - 0-55 (per physician preference for patients over 6) ATG/Flu/Bu
  Interventions: Biological: Cell Infusion; Drug: Thymoglobulin; Drug: Fludarabine; Drug: Busulfan; Drug: Tacrolimus; Drug: Mycophenolate Mofetil
- Arm C (Experimental): Arm C Fully Matched unrelated donor (MUD)- - 0-55 years; ATG/Flu/Bu
  Interventions: Biological: Cell Infusion; Drug: Thymoglobulin; Drug: Fludarabine; Drug: Busulfan; Drug: Tacrolimus; Drug: Mycophenolate Mofetil
- Arm D (Experimental): Arm D: Haploindentical or mismatched unrelated donors (MMUD) - 0-55 years; ATG/Thiotepa/Cyclophosphamide/MESNA/Flu/TBI
  Interventions: Radiation: Total Body Irradiation; Biological: Cell Infusion; Drug: Thymoglobulin; Drug: Fludarabine; Drug: Thiotepa; Drug: Cyclophosphamide; Drug: Sirolimus; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab (Campath) will be administered IV over 2 hours on day -8 to day -4.
  Other Names: Campath
  Arms: Arm A
Radiation: Total Body Irradiation — 400 cGy in 2 split fractions will be administered per Department of RadiationOncology SOPs.
  Other Names: TBI
  Arms: Arm A; Arm D
Biological: Cell Infusion — On day 0 the cells will be infused per cell source specific institutional guidelines
Drug: Thymoglobulin — ATG will be administered IV every 24 hours beginning on day -8 for all patients.
  Dosing will be model-based using Bayesian methodology13,14,15. Total doses and total number of doses (1-4 doses) will be determined based on absolute lymphocyte count and weight.
  Other Names: Rabbit ATG
  Arms: Arm B; Arm C; Arm D
Drug: Fludarabine — Fludarabine will be administered IV over 1 hour every 24 hours on day -5 to day - 2. The daily dose of fludarabine will be determined by model-based dosing utilizing Bayesian methodology with a cumulative area under the curve (cAUC) of 20 mg*hr/L (range 18-22 mg*hr/L).
  Arms: Arm B; Arm C; Arm D
Drug: Busulfan — Busulfan dosing and administration and therapeutic drug monitoring (TDM) per institutional guidelines. Initial busulfan dosing will be determined by model-based dosing utilizing Bayesian methods with a cumulative area under the curve (cAUC) of 75 mg*hr/L.
  Arms: Arm B; Arm C
Drug: Thiotepa — Thiotepa will be administered at a dose 5 mg/kg IV every 12 hours on day - 7 over 2 hours. Patients will undergo thiotepa skin care per institutional guidelines
  Arms: Arm D
Drug: Cyclophosphamide — Cyclophosphamide will be administered at a dose of 14.5 mg/kg over 2 hours IV daily on days -6 and -5. Cyclophosphamide dosing is calculated based on actual body weight (ABW).
  For Arm D - Cyclophosphamide 50 mg/kg IV will be administered over 2 hours on days +3 and
  +4. Cyclophosphamide dosing for post-transplant is calculated based on ideal body weight (IBW) unless patient weighs less than IBW, in which case actual body weight (ABW) will be used.
  Other Names: Cyclophosphamide with MESNA
  Arms: Arm D
Drug: Sirolimus — Patients on Arm A and Arm D will receive sirolimus; beginning on day -3 and continuing until day +180 for patients on Arm A or beginning on day +5 and continuing until 1 year post transplant for patients on Arm D.
  Arms: Arm A; Arm D
Drug: Tacrolimus — Patients on Arm B and Arm C will receive tacrolimus, beginning on day -3 and continuing until day +180. Tacrolimus dosing and monitoring will be per institutional guidelines.
  Arms: Arm B; Arm C
Drug: Mycophenolate Mofetil — MMF will begin on day -3 (Arm A, B & C) or day +5 (Arm D). Patients treated on adult service will receive 15 mg/kg (max 1500 mg/dose) given every 12 hours, rounded to nearest 250 mg. Patients on pediatric service will receive 15 mg/kg (max 1000 mg/dose) given every 8 hours. MMF dosing will be monitored and altered as clinically appropriate based on institutional guidelines. MMF will be stopped at day +30 (Arms A, B & C) or day +35 (Arm D) or 7 days after engraftment, whichever day is later, if no acute GVHD.
  Other Names: (MMF)

SUMMARY:
A single center, open label, interventional, phase II trial for donor transplant for high risk hemoglobinopathies and other red cell transfusion dependent disorders utilizing allogeneic hematopoietic stem cell transplantation (HSCT) regimens.

ELIGIBILITY:
Inclusion Criteria:

* Sickle Cell Disease (SCD)
* SCD Patients with a fully matched sibling donor (MSD) irrespective of the frequency or severity of symptoms MSD transplant can be considered. Parents/patient must be counseled as to the risks and benefits and provide their voluntary informed consent
* Transfusion Dependent Alpha- or Beta- Thalassemia
* Diamond Blackfan Anemia
* Other Non-Malignant Hematologic Disorders
* Karnofsky ≥ 60%, Lansky play score ≥ 60. Patients with lower performance score can be considered based on study team's evaluation.
* Sexually active persons of childbearing potential or persons with partners of childbearing potential must agree to use a highly effective form of contraception during study treatment and for at least 4 months after the transplant.

Exclusion Criteria:

* Pregnant, breastfeeding or intending to become pregnant during the study. Persons of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days of the start of treatment
* HIV Positive
* Active, uncontrolled infection - infection that is stable or improving after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections) will be permitted
* Known allergy to any of the study components
* Psychiatric illness/social situations that, in the judgement of the enrolling Investigator, would limit compliance with study requirements
* Other illness or a medical issue that, in the judgement of the enrolling Investigator, would exclude the patient from participating in this study

Max Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Graft versus Host Disease (GvHD) | 1 year

SECONDARY OUTCOMES:
Overall Survival | 1 and 2 years
  Overall survival post HCT
Grade 3-4 Acute GvHD | 2 years
  Grade 3-4 acute Graft versus Host Disease (GvHD) at 2 years post HCT.
Chronic Graft versus Host Disease (GvHD) Free | 2 years
  Chronic Graft versus Host Disease (GvHD) Free at 2 years post HCT.
Failure Free Survival | 2 years
  Failure Free Survival 2 years post HCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States